CLINICAL TRIAL: NCT05190263
Title: Quality Assurance on Anemia Management in Patients With Solid Tumors and Malignant Lymphoma
Acronym: QA Anemia
Status: Completed | Type: Observational
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Prof. Hartmut Link (Unknown); MMF GmbH (Industry); AIO AG Supportivtherapie (Other); AG Supportive Maßnahmen in der Onkologie (Other)
Responsible Party: Sponsor
Other Study IDs: AIO-SUP-0121
Record Dates: First submitted 2021-12-14; First posted 2022-01-13 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Anemia, Iron Deficiency; Solid Tumor; Malignant Lymphoma
MeSH Terms: conditions — Anemia, Iron-Deficiency; Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-interventional retrospective epidemiological observational study — non-interventional retrospective epidemiological observational study

SUMMARY:
The aim of the study is to analyze the implementation of the 2018 updated ESMO Guideline in patients with tumor diseases as well as the corre-sponding recommendations of the Onkopedia Guideline and the S3 Guide-line Supportive Therapy in routine clinical practice in Germany.

To this end, a nationwide, representative, retrospective patient documen-tation will be conducted to observe the current practice of anemia man-agement in hospitals and among office-based physicians.

DETAILED DESCRIPTION:
Health care structure analysis and recruitment (phase 1):

In a first step, data on care facilities treating patients in the above indica-tions in Germany will be collected (gastroenterology, gynecology, hema-tology/oncology, and pneumology hospital departments, as well as of-fice-based hematologists/oncologists and gynecology oncologists).

In Phase 1, all centers in Germany potentially treating patients in the above entities will be contacted and data on the care level of the institu-tion and the number of patients treated will be collected using a one-page pen-to-paper form. In addition, the willingness of the care facilities to participate in the documentation of patients will be surveyed (Phase 2).

Analysis of patient records (phase 2)

In order to obtain a reliable, representative sample of patients treated in Germany, the distribution of the cases to be documented in the individual indications among the participating facilities is determined. For this pur-pose, the data collected from the facilities in Phase I on patient numbers and treatment structure will be used:

Participating centers are divided into clusters based on key distinguishing characteristics (facility type, level of care, and number of patients treat-ed). This sample is modulated according to the previous care structure analysis. This approach allows the actual percentages of the different care facilities in an indication area to be proportionally included in the patient documentation sample.

In Phase 2, a multi-page electronic case record form (eCRF) will be com-pleted to collect patient and treatment data relevant to the purpose of the study. All data will be collected retrospectively and anonymously from patient records.

* Patient- and disease-related variables (age, ECOG performance status, staging, relevant comorbidities).
* Drug therapy (chemotherapy, antibodies, immunotherapy, kinase inhibitors: Start/end, substances or regimens).
* Radiotherapy (start/end, irradiated region)
* Laboratory diagnostics (if available) with Hb, Hk, MCV, MCH, re-ticulocytes and/or Ret-Hb, ferritin, transferrin and/or transferrin saturation (TSAT), holo-trans-cobalamin (vitamin B12), folic acid, zinc protoporphyrin, creatinine clearance (GFR), EPO level
* Data on anemia therapy (transfusion of RBC; iron therapy p.o. or i.v.; ESA). To ensure data quality, the scientific project lead will train two employees of the commissioned institute in content-related issues of the study. This knowledge will be incorporated into the programming of the user inter-face and the patient databases so that the program will check for com-pleteness and, as far as possible, plausibility based on defined require-ments and framework conditions. These checks accompany the process of data entry into the eCRF and enable immediate validation of the data.

ELIGIBILITY:
Inclusion Criteria:

Patients

* with antineoplastic therapy (chemotherapy or "new substances"), radiochemotherapy or radiotherapy in the period 1/1/2021 - 06/30/2021
* with anemia with hemoglobin levels decreases below 10g/dl (6.2 mmol/l) at least once during the period 1/1/2021 - 06/30/2021
* with at least 4 weeks of follow up period after anemia diagnosis.

Exclusion Criteria:

* Follow up time less than 4 weeks,
* lack of patient contact after anemia diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors or malignant lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
See result section upon availability | 06/2021 - 09/2022
  The ESMO Guideline "Management of Anemia and Iron Deficiency in Patients with Cancer", updated in 2018, provides a dedicated algorithm to guide decision-making in the diagnosis and treatment of anemia in tumor patients in order to reduce anemia-related complications. This includes recommendations on
  * iron therapy,
  * erythropoiesis stimulating agents (ESA) and
  * transfusion with red blood cells (RBC) depending on various diagnostic parameters and the respective antitumor therapy. The therapy recommendations presented correspond with the recommendations of the Onkopedia guideline on iron deficiency anemia, the S3 guideline on supportive therapy and the cross-sectional guidelines for therapy with blood components and plasma derivatives.
  To this end, this study examines the common practice of adherence to the algorithm of guideline adherence by reviewing the above criteria such as iron therapy, use of ESA and RBC substitution.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Link, Prof. Dr., Principal Investigator — AIO AG Supportive Therapie
Locations (1):
- Studienzentrum Prof. Dr. med. Hartmut Link, Facharzt für Innere Medizin, Hämatologie und Internistische Onkologie, Kaiserslautern, Germany

IPD SHARING:
Plan to Share IPD: No
Data is collected retrospectively and completely anonymously from patient records, no identifying characteris-tics (e.g. birth date, initial letters, pseudonym) will be collected.
  It is hoped that these data will assist in creating new possibilities and ways to improve the quality of treatment through further training and enhancement of the availability and transparency of the guidelines.

REFERENCES:
- [Derived] Link H, Kerkmann M, Holtmann L, Detzner M. Anemia diagnosis and therapy in malignant diseases: implementation of guidelines-a representative study. Support Care Cancer. 2024 Jan 19;32(2):113. doi: 10.1007/s00520-023-08267-4. PMID 38240843